CLINICAL TRIAL: NCT01914926
Title: DiME Study: Comparison of Diltiazem and Metoprolol in the Management of Acute Atrial Fibrillation or Atrial Flutter With Rapid Ventricular Response: A Prospective Randomized and Double-Blinded Non-Inferiority Trial of Safety and Efficacy
Brief Title: Comparison of Diltiazem and Metoprolol in the Management of Acute Atrial Fibrillation or Atrial Flutter
Acronym: DiME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09/01/VA02
Record Dates: First submitted 2013-07-11; First posted 2013-08-02 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Heart Rate and Rhythm Disorders
Keywords: metoprolol; diltiazem; heart rate
MeSH Terms: interventions — Metoprolol; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoprolol Study Group (Active Comparator): Patients Receiving metoprolol administered at a dose of 0.15 mg/kg (to a maximum dose of 10 mg)
  Interventions: Drug: Metoprolol
- Diltiazem Study Group (Active Comparator): Patients receiving diltiazem administered parenterally at a dose of 0.25 mg/kg (to a maximum dose of 30 mg)
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Metoprolol
  Arms: Metoprolol Study Group
Drug: Diltiazem
  Arms: Diltiazem Study Group

SUMMARY:
Acute atrial fibrillation is the most common sustained, clinically significant dysrhythmia encountered in the emergency department (ED) and the most common dysrhythmia treated by emergency physicians. Atrial flutter is less common than atrial fibrillation but its management in the ED is very similar, and the majority of patients with atrial flutter also have atrial fibrillation. Symptomatic relief and ventricular rate control are generally the primary therapeutic objectives in the ED management of acute atrial fibrillation and flutter (AFF). The need for swift, appropriate action by the emergency physician is highlighted by the fact that up to 18% of patients with AFF develop potentially life-threatening complications such as congestive heart failure, hypotension, ventricular ectopy, respiratory failure, angina and myocardial infarction.

Both beta-blocking agents and calcium channel blockers are commonly used to treat AFF in the ED. Metoprolol is the most commonly used beta-blocker; and diltiazem is the most frequently used calcium channel antagonist.[8] Diltiazem was released by the FDA for treatment of AFF in 1992. Shreck et al. were the first to demonstrate both the efficacy of diltiazem in the ED management of AFF with rapid rate and its clear superiority over the previously most commonly used pharmacologic agent, digoxin.

To date, only one prospective, randomized trial has compared the effectiveness of a calcium channel blocker (diltiazem) with a beta-blocker (metoprolol) for rate control of AFF in the ED. Despite the relatively small sample size (n=20 in each group) the authors concluded that both pharmacologic agents were similarly effective. In order to test this finding, the investigators conducted a prospective comparison of metoprolol and diltiazem for the management of patients presenting to the ED with AFF with rapid ventricular rate.

DETAILED DESCRIPTION:
We conducted a prospective, randomized, double-blind study to compare the effectiveness of intravenous metoprolol with that of diltiazem in achieving rate control in adult ED patients with rapid atrial fibrillation or flutter. Approval of the study was obtained from our hospital's institutional review board. All enrolled patients provided written informed consent and HIPAA authorization documentation.

This study was set in the adult ED of Maimonides Medical Center, an urban teaching hospital in Brooklyn, NY with an annual ED census of more than 120,00 patients. A convenience sample of adult patients age 18 or older presenting with a supraventricular tachydysrhythmia were evaluated for enrollment. Eligible patients had to have a 12-lead electrocardiogram (ECG) showing atrial fibrillation or atrial flutter with a ventricular rate of greater than or equal to 120 beats per minute. Data collected included demographics, medical history, vital signs and electrocardiogram findings. All patients were immediately evaluated by the treating physician utilizing ACLS protocols. At the discretion of the treating physician, intravenous adenosine was administered in order to facilitate identification of the underlying supraventricular tachydysrhythmia. All patients were attached to a monitor that displays cardiac rhythm, heart rate, blood pressure and oxygen saturation.

Upon enrollment, patients were randomly assigned, in a 1:1 ratio, to receive diltiazem administered parenterally at a dose of 0.25 mg/kg (to a maximum dose of 30 mg) or metoprolol administered at a dose of 0.15 mg/kg (to a maximum dose of 10 mg). Randomization was performed through the use of a computer-generated randomization list. Pharmacy released the study drug in a locked tackle box coded in number sequence to correspond to that of the computer-generated randomization list, upon which the pharmacist also prepared the study drug in blinded fashion. The study medications were packaged in identical-appearing dispensing kits. Patients who were randomly assigned to diltiazem received a bolus injection in a syringe that appeared identical to that of metoprolol. Admixture and labeling were performed by the pharmacist in the ED and dispensed to the treating nurse for administration. Doses of each study medication were adjusted with normal saline to a total of 10 ml in each syringe to prevent un-blinding. The time at which the first dose was administered was denoted as time zero (baseline). If the primary endpoint was not achieved at time 15 minutes, then a second escalation dose was administered. If the patient had been enrolled in the diltiazem group, the escalation dose was 0.35 mg/kg (to a maximum dose of 30 mg), and for patients enrolled in the metoprolol group, the escalation dose was 0.25 mg/kg (to a maximum dose of 10 mg). As with the initial dose, the escalation dose was prepared by the pharmacist and given to the treating nurse for patient administration in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients had to have a 12-lead electrocardiogram (ECG) showing atrial fibrillation or atrial flutter with a ventricular rate of greater than or equal to 120 beats per minute and a systolic blood pressure of greater than or equal to 90 mmHg.

Exclusion Criteria:

Patients were excluded if they had any of the following:

* a systolic blood pressure <90 mmHg, ventricular rate greater than or equal to 220 beats per minute,
* QRS >0.100 seconds, 2nd or 3rd degree atrioventricular (AV) block,
* temperature >38.0 ˚C,
* acute ST elevation myocardial infarction,
* known history of New York Heart Association Class IV heart failure or
* active wheezing with a history of bronchial asthma or COPD.

In addition, patients were excluded if there was:

* prehospital administration of diltiazem or any other AV nodal blockading agent,
* a history of cocaine or methamphetamine use in the previous 24 hours prior to arrival,
* a history of allergic reaction to diltiazem or metoprolol,
* a history of sick sinus or pre-excitation syndromes,
* a history of anemia with hemoglobin <11.0 g/dl,
* pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Study Chair — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Scott PA, Pancioli AM, Davis LA, Frederiksen SM, Eckman J. Prevalence of atrial fibrillation and antithrombotic prophylaxis in emergency department patients. Stroke. 2002 Nov;33(11):2664-9. doi: 10.1161/01.str.0000035260.70403.88. PMID 12411658
- [Background] McDonald AJ, Pelletier AJ, Ellinor PT, Camargo CA Jr. Increasing US emergency department visit rates and subsequent hospital admissions for atrial fibrillation from 1993 to 2004. Ann Emerg Med. 2008 Jan;51(1):58-65. doi: 10.1016/j.annemergmed.2007.03.007. Epub 2007 Apr 27. PMID 17466409
- [Background] Friberg J, Buch P, Scharling H, Gadsbphioll N, Jensen GB. Rising rates of hospital admissions for atrial fibrillation. Epidemiology. 2003 Nov;14(6):666-72. doi: 10.1097/01.ede.0000091649.26364.c0. PMID 14569181
- [Background] Wattigney WA, Mensah GA, Croft JB. Increasing trends in hospitalization for atrial fibrillation in the United States, 1985 through 1999: implications for primary prevention. Circulation. 2003 Aug 12;108(6):711-6. doi: 10.1161/01.CIR.0000083722.42033.0A. Epub 2003 Jul 28. PMID 12885749
- [Background] Stiell IG, Clement CM, Perry JJ, Vaillancourt C, Symington C, Dickinson G, Birnie D, Green MS. Association of the Ottawa Aggressive Protocol with rapid discharge of emergency department patients with recent-onset atrial fibrillation or flutter. CJEM. 2010 May;12(3):181-91. doi: 10.1017/s1481803500012227. PMID 20522282
- [Background] Friedman HZ, Goldberg SF, Bonema JD, Cragg DR, Hauser AM. Acute complications associated with new-onset atrial fibrillation. Am J Cardiol. 1991 Feb 15;67(5):437-9. doi: 10.1016/0002-9149(91)90059-t. No abstract available. PMID 1994672
- [Background] Chenoweth J, Diercks DB. Management of atrial fibrillation in the acute setting. Curr Opin Crit Care. 2012 Aug;18(4):333-40. doi: 10.1097/MCC.0b013e328354dc30. PMID 22622515
- [Background] Demircan C, Cikriklar HI, Engindeniz Z, Cebicci H, Atar N, Guler V, Unlu EO, Ozdemir B. Comparison of the effectiveness of intravenous diltiazem and metoprolol in the management of rapid ventricular rate in atrial fibrillation. Emerg Med J. 2005 Jun;22(6):411-4. doi: 10.1136/emj.2003.012047. PMID 15911947
- [Background] Kovacic JC, Moreno P, Nabel EG, Hachinski V, Fuster V. Cellular senescence, vascular disease, and aging: part 2 of a 2-part review: clinical vascular disease in the elderly. Circulation. 2011 May 3;123(17):1900-10. doi: 10.1161/CIRCULATIONAHA.110.009118. No abstract available. PMID 21537006
- [Background] Stiell IG, Macle L; CCS Atrial Fibrillation Guidelines Committee. Canadian Cardiovascular Society atrial fibrillation guidelines 2010: management of recent-onset atrial fibrillation and flutter in the emergency department. Can J Cardiol. 2011 Jan-Feb;27(1):38-46. doi: 10.1016/j.cjca.2010.11.014. PMID 21329861
- [Background] Rogenstein C, Kelly AM, Mason S, Schneider S, Lang E, Clement CM, Stiell IG. An international view of how recent-onset atrial fibrillation is treated in the emergency department. Acad Emerg Med. 2012 Nov;19(11):1255-60. doi: 10.1111/acem.12016. PMID 23167856
- [Background] Maxwell CJ, Hogan DB, Campbell NR, Ebly EM. Nifedipine and mortality risk in the elderly: relevance of drug formulation, dose and duration. Pharmacoepidemiol Drug Saf. 2000 Jan;9(1):11-23. doi: 10.1002/(SICI)1099-1557(200001/02)9:13.0.CO;2-U. PMID 19025798
- [Background] Jollis JG, Simpson RJ Jr, Chowdhury MK, Cascio WE, Crouse JR 3rd, Massing MW, Smith SC Jr. Calcium channel blockers and mortality in elderly patients with myocardial infarction. Arch Intern Med. 1999 Oct 25;159(19):2341-8. doi: 10.1001/archinte.159.19.2341. PMID 10547174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients was from June 2009 to November 2010
Pre-assignment Details: No significant events
Period: Overall Study
Arm/Group | Metoprolol Study Group | Diltiazem Study Group
Started | 29 | 25
Completed | 28 | 24
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — uncooperative, agitated and removed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoprolol Study Group | Diltiazem Study Group | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 18 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.95 (14.94) | 65.85 (13.22) | 67.52 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 29 | 25 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Reaching Target HR<100bpm Within 30 Minutes
Description: Percent of patient who reached a HR<100bpm within 30 minutes from baseline.
Time Frame: 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Metoprolol Study Group | Diltiazem Study Group
Number analyzed (Participants) | 28 | 24
percentage of participants | 46.4 | 95.8
Statistical Analysis 1: Comparison: Metoprolol Study Group vs Diltiazem Study Group; We estimated a sample size of 200 patients assigned in a 1:1 ratio to receive diltiazem and metoprolol would achieve 80% power to detect non-inferiority using a one-sided two sample t-test. The margin of equivalence is -10; Test type: Non-Inferiority or Equivalence — Chi-Square test; p = .0001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Metoprolol Study Group | Diltiazem Study Group
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes